CLINICAL TRIAL: NCT02764697
Title: Prospective Open Label Study of H.P. Acthar Gel Injection in Patients With Active Non-Infectious Uveitis With Associated Glaucoma Thus High Frequency Regional Corticosteroid and Oral Corticosteroids Cause Intolerable Side-Effects
Brief Title: Study of H.P. ACTHAR Subcutaneous Gelatin (Gel)(Highly Purified Gel Injection) in Uveitis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampa Bay Uveitis Center, LLC (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBUC 10012015
Record Dates: First submitted 2016-04-25; First posted 2016-05-06 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Uveitis; Anterior Uveitis; Intermediate Uveitis; Posterior Uveitis; Scleritis; Clinically Significant Macular Edema
Keywords: Glaucoma associated with uveitis
MeSH Terms: conditions — Uveitis; Uveitis, Anterior; Uveitis, Intermediate; Uveitis, Posterior; Scleritis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- H.P. Acthar Subcutaneous Gel Injection (Other): For the current protocol we are proposing, 40 U/ml, given twice weekly x 8 weeks, followed by once weekly x 4 weeks: a total 20 doses, using the approved route, with the option to do 4 additional doses if resolution is incomplete.
  Interventions: Drug: H.P. ACTHAR SUBCUTANEOUS GEL INJECTION

INTERVENTIONS:
Drug: H.P. ACTHAR SUBCUTANEOUS GEL INJECTION — Subcutaneous injection twice weekly
  Other Names: Acthar

SUMMARY:
Uveitis represents a heterogeneous group of diseases that results from ocular inflammatory reaction involving ocular tissue and vasculature. The inflammation usually causes pain, redness, photophobia and blurred vision. This inflammation, is typically treated with regional or systemic therapy. The regional therapy typically consists of topical corticosteroids or periocular or regional corticosteroids. Regional therapy can lead to a steroid response glaucoma, which is increased intraocular pressure.This pilot study aims to evaluate the possible effectiveness of H.P. Acthar in patients with active ocular inflammatory disease, and currently on treatment for glaucoma or have a history of glaucoma.

DETAILED DESCRIPTION:
Uveitis represents a heterogeneous group of diseases that results from ocular inflammatory reaction involving ocular tissue and vasculature. The inflammation usually causes pain, redness, photophobia and blurred vision.

H.P Acthar Gel stimulate the adrenal cortex to secrete cortisol. Additionally H.P. Acthar gel is also reported to bind to melanocortin receptors. Melanocortin receptor activation has been shown to exert marked anti-inflammatory and immune-modulatory effects in animal studies, by modulating pro inflammatory cytokines, followed by induction of anti- inflammatory mediators and subsequent leukocyte migration. Specifically melanocortins down regulate Tumor Necrosis Factor (TNF) alpha, Interleukin (IL) -2, Interferon gamma and T-cell proliferation and upregulates IL-10 and regulatory T cells. For this reason H.P. Acthar is an approved treatment for ocular inflammatory disease.

Ocular inflammatory disease is typically treated with regional or systemic therapy. The regional therapy typically consists of topical corticosteroids or periocular or regional corticosteroids. Regional therapy can lead to a steroid response glaucoma, which is increased intraocular pressure.This pilot study aims to evaluate the possible effectiveness of H.P. Acthar in patients with active ocular inflammatory disease, and currently on treatment for glaucoma or have a history of glaucoma.

Subjects will be treated with H P Acthar subcutaneous gel, 40 U/ml, given twice weekly x 8 weeks, followed by once weekly x 4 weeks: a total 20 doses with the same cumulative units to be administered, using the approved route, with the option to do 4 additional doses if resolution is incomplete.

This will be a prospective open-label, non-randomized pilot study: 12 week treatment for active non-infectious uveitis, endpoint assessment and safety assessment; additional 12 week assessment for uveitis activity/quiescence and safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Subject has the ability to understand and sign the informed consent document
* Subject is 18 years of age or older
* Subject can be male or female
* Subject has negative Purified Protein Derivative (Tuberculosis skin test) or quantiferon TB Gold Test (blood test for TB) testing done in 3 months
* Subject has active ocular inflammation in at least one eye
* Subject has visual acuity in at least one eye of 20/400 or better.
* Subject has a history of glaucoma or has actively treated glaucoma
* Subject is willing and able to comply with the study procedures
* Female subjects of childbearing potential must not be pregnant or breast-feeding, must have a negative pregnancy test at screening and must be willing to undergo pregnancy testing throughout the study

Exclusion Criteria:

* Subject has any ocular infection
* Subject has any systemic infection
* Participant has documented immunocompromised or immune-incompetent state
* Subject has any ocular co-morbidity than prevents assessment of intraocular inflammation
* Subject has had any intra-ocular surgery in previous 6 weeks
* Subject has any planned elective surgery ocular or systemic during study duration
* Subject is pregnant or breast-feeding
* Subject had a recent vaccination with live or attenuated vaccines
* Subject has a sensitivity to Porcine derived proteins
* Subject has a medical history which is a contraindication to receiving H.P. Acthar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2016-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace L Clarke, Principal Investigator — Tampa Bay Uveitis Center, LLC
Locations (1):
- Tampa Bay Uveitis Center, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was 06/31/2016 through 08/10/2016
  Active follow-up period 06/31/2016 through 12/07/2016
  The study was conducted at 1 site Tampa Bay Uveitis Center, LLC 5800 49th Street North, St Petersburg Fl 33709: Outpatient Medical Clinic
Pre-assignment Details: The patient after consent was given, were required to have their medical records reviewed and have screening laboratory evaluations
Period: Overall Study
Arm/Group | H.P. Acthar Subcutaneous Gel Injection
Started | 5
Completed | 2
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | H.P. Acthar Subcutaneous Gel Injection
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Photographic Haze Reduced to Grade 0 or Down 2 Steps Documented With Fundus Photography
Description: Subjects will have fundus photography at baseline and 12 weeks. Intermediate uveitis is graded by haze; it is done using the photographic scale: grades 0-4 (lower values are a better outcome), utilized by the SUN criteria, based on the Nussenblatt photographic vitreous haze scale
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | H.P. Acthar Subcutaneous Gel Injection
Number analyzed (Participants) | 5
Participants
  1 Step of VH Improvement | 3
  2 Step of VH | 1
  No VH Improvement | 1

2. Primary Outcome: Number of Participants With Clinically Significant Improvement of Macular Edema
Description: Clinically Significant Uveitic Macular Edema: Clinical Improvement of Macular Edema with OCT Documentation of central foveal thickness < 300 microns
Time Frame: 12 weeks
Population: 0
Measure: Count of Participants; unit: Participants
Arm/Group | H.P. Acthar Subcutaneous Gel Injection
Number analyzed (Participants) | 5
Participants
  Decrease in Central Foveal Thickness <300 | 0
  Decrease in central Fovea > 300 Microns | 5

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | H.P. Acthar Subcutaneous Gel Injection
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No